CLINICAL TRIAL: NCT02592928
Title: Regional Implementation of Collaborative Lung Function Testing
Acronym: e-Spiro-HC3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government); Fundació TicSalut (Other); Institut Catala de Salut (Other Government); Fundació Eurecat (Other); Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Felip Burgos, PhD, RN, Hospital Clinic of Barcelona
Other Study IDs: 2015-PDMAR
Record Dates: First submitted 2015-10-15; First posted 2015-10-30 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Integrated Care; Telehealth; Health Care Rationing
Keywords: eHealth; Spirometry; Lung Function; Primary Care; Telehealth; Integrated Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lleida Health Sector: Lleida (168k inhabitants and 21 Primary Care centers). Primary Care centers from this health sector
  Inclusion of the Forced Spirometry into the Electronic Health Records No interventions performed
  Interventions: Other: Inclusion of Spirometry into the Electronic Health Records
- Vic Health Sector: Vic (49k inhabitants and 11 Primary Care Centers). Primary Care centers from this health sector
  Inclusion of the Forced Spirometry into the Electronic Health Records No interventions performed
  Interventions: Other: Inclusion of Spirometry into the Electronic Health Records
- AISBE Health Sector: Atenció Integral en Salut Barcelona Esquerra (AISBE) (540k inhabitants and 19 Primary Care centers). Primary Care centers from this health sector
  Inclusion of the Forced Spirometry into the Electronic Health Records No interventions performed
  Interventions: Other: Inclusion of Spirometry into the Electronic Health Records

INTERVENTIONS:
Other: Inclusion of Spirometry into the Electronic Health Records — Inclusion of the Forced Spirometry into the Electronic Health Records
  Other Names: Follow up using Plan-Do-Study-Act (PDSA) methodology

SUMMARY:
Background/Aims There is evidence indicating that deployment of forced spirometry (FS) testing in a collaborative scenario, encompassing respiratory specialists and community professionals, generates healthcare efficiencies. The study describes the roadmap for regional implementation of the FS program in Catalonia (ES), from January to December 2016.

Methods/Design Firstly, the FS program will be deployed in three healthcare sectors (514 k inhabitants), following Plan-Do-Study-Act iterative cycles, using the Model for Assessment of Telemedicine for evaluation purposes. Thereafter, regional deployment of the FS program (7.5M inhabitants) will be conducted. The third step considers: evaluation of transferability, preparation for data analytics and recommendations for long-term assessment of outcomes. Main components of the FS program are: i) Automatic quality testing; ii) Standardized data transfer to a shared electronic health record; iii) Elaboration of individual FS reports including historical results; and, iv) Clinical decision support systems providing access to the FS report, and to remote support upon request.

Discussion/Conclusions The project constitutes the first attempt to scale-up a collaborative scenario for FS testing that will open new avenues for longitudinal lung function assessment. Moreover, the setting shows high potential for transferability to different sites and to other diagnostic procedures.

DETAILED DESCRIPTION:
The Forced Spirometry program emerges from a series of studies reporting on technological solutions for each of the main components indicating the potential of their articulated application aiming at covering unmet needs for collaborative FS testing. The studies were initiated within the EU project NEXES22;23 and specific parts of the overall setting have already been successfully evaluated in the Basque Country.

The setting & Study design The current protocol has been designed as part of the regional deployment of integrated care services in Catalonia. It consists of the two lines of activity ultimately aiming at: i) regional adoption of the FS program; and, ii) generalization of the approach to other areas, as well as to other testing procedures. The research was submitted and apoved by the Ethical Committee of the Hospital Clínic i Provincial de Barcelona.

Program deployment The initial 6 months will include three healthcare sectors: Lleida (168k inhabitants and 21 Primary Care centers), Vic (49k inhabitants and 11 PCC), and Atenció Integral en Salut Barcelona Esquerra (AISBE) (540k inhabitants and 19 PCC) following a Plan-Do-Study-Act (PDSA) methodology24. The first PDSA cycle (January - March 2016) including a total of three primary care centers, one in each healthcare sector, has as main purpose to ensure full functionality of the setting. Immediately thereafter, the FS program will be progressively deployed to all Primary Care centers in the three sectors in a second 3-months PDSA cycle that will be completed by mid-2016. Forced spirometry testing will be prescribed by the attending general practitioner following standard criteria and it will be carried out by primary care nurses.

The deployment of the program in the entire region (7.5M inhabitants and 369 Primary Care centers) will be completed with no discontinuation within 2016. It will follow identical PDSA methodology. The outcomes of the assessment carried out during each PDSA cycle will modulate the long-term assessment strategy of the FS program described below.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the regular practice

Exclusion Criteria:

* Clinical an Medical exclusion criteria as the forced spirometry standards recommend.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The initial 6 months will include 3 healthcare sectors: Lleida (168k inhabitants, 21 Primary Care Centers), Vic (49k inhabitants, 11 PCC), and AISBE (540k inhabitants, 19 PCC) following a Plan-Do-Study-Act (PDSA) methodology. The first PDSA cycle (January - March 2016) including a total of 3 PCC, one in each healthcare sector, has as main purpose to ensure full functionality of the setting. The FS program will be progressively deployed to all PCC in the 3 sectors in a second 3-months PDSA cycle that will be completed by mid-2016. FS testing will be prescribed by general practitioner following standard criteria and it will be carried out by primary care nurses. The deployment in the entire region (7.5M inhabitants and 369 Primary Care centers) will be completed within 2016.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of Primary Care Centers (PCC) and professionals involved in the territory using the Electronic Health Records (EHR) | Thought study completition in average of 18 months
  Number of PCC exporting both the raw spirometric data, including all FS curves, and the FS report to the shared electronic health record at a regional level.
Number of professionals using Forced Spirometry included in the EHR (percentage per PCC) | Thought study completition in average of 18 months
  Number of professionals with accessi of the FS testing report, irrespective of the healthcare provider and health level wherein testing was performed
Change between inicial and end of the project (number of FS test included in the EHR) | Thought study completition in average of 18 months

SECONDARY OUTCOMES:
Forced Spirometry Parameters | Thought study completition in average of 18 months
  - Measured in liters
Grade of quality in relation of total Forced Spirometry | Thought study completition in average of 18 months
  Percentage of patients with FS grade of quality (A-B-C-D-F) in relation of total FS
Change from baseline in relations with ascertainment of COPD or Asthma diagnosis | Thought study completition in average of 18 months
  * Percentage of patients with FEV1/FVC ratio < 0.7 and without diagnosis of Asthma and COPD
  * Percentage of patients with FEV1/FVC ratio > 0.7 and with diagnosis Asthma and COPD
  * Percentage of patients with restrictive pattern and FEV1/FVC ratio < 0.7
Number of participants per PCC | Through study completion, an average of 18 months
  Long-term benefits from data analytics of longitudinal information
  Assessments using unique measurements
Grade of satisfaction about new servicies | Through study completion, an average of 18 months
  Grade of satisfaction about new servicies (0-10)
Rating the degree of clinical impact to obtain the historical spirometry values of each patient. | Through study completion, an average of 18 months
  Rating the degree of clinical impact to obtain the historical spirometry values of each patient. Grade 0 -10
Number of avoided duplication tests using the EHR | Through study completion, an average of 18 months
  Number of avoided duplication tests using the EHR. measured as % of the total FS
Cost-effectiveness (Rating usability and speed of data transfer) | Through study completion, an average of 18 months
  Rating usability and speed of data transfer in minutes .
Cost-effectiveness (reducing the time of access to information and better display of the information) | Through study completion, an average of 18 months
  Questionnaire about reducing the time of access to information and better display of the information (measured in minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Felip Burgos, Barcelona, Spain

REFERENCES:
- [Background] Cano I, Alonso A, Hernandez C, Burgos F, Barberan-Garcia A, Roldan J, Roca J. An adaptive case management system to support integrated care services: Lessons learned from the NEXES project. J Biomed Inform. 2015 Jun;55:11-22. doi: 10.1016/j.jbi.2015.02.011. Epub 2015 Mar 18. PMID 25796455
- [Background] Burgos F, Melia U, Vallverdu M, Velickovski F, Lluch-Ariet M, Caminal P, Roca J. Clinical decision support system to enhance quality control of spirometry using information and communication technologies. JMIR Med Inform. 2014 Oct 21;2(2):e29. doi: 10.2196/medinform.3179. PMID 25600957
- [Background] Melia U, Burgos F, Vallverdu M, Velickovski F, Lluch-Ariet M, Roca J, Caminal P. Algorithm for automatic forced spirometry quality assessment: technological developments. PLoS One. 2014 Dec 31;9(12):e116238. doi: 10.1371/journal.pone.0116238. eCollection 2014. PMID 25551213
- [Background] Velickovski F, Ceccaroni L, Roca J, Burgos F, Galdiz JB, Marina N, Lluch-Ariet M. Clinical Decision Support Systems (CDSS) for preventive management of COPD patients. J Transl Med. 2014 Nov 28;12 Suppl 2(Suppl 2):S9. doi: 10.1186/1479-5876-12-S2-S9. Epub 2014 Nov 28. PMID 25471545
- [Background] Llauger MA, Rosas A, Burgos F, Torrente E, Tresserras R, Escarrabill J; en nombre del grupo de trabajo de espirometria del Plan Director de las Enfermedades del Aparato Respiratorio (PDMAR). [Accesibility and use of spirometry in primary care centers in Catalonia]. Aten Primaria. 2014 Jun-Jul;46(6):298-306. doi: 10.1016/j.aprim.2013.12.012. Epub 2014 Apr 24. Spanish. PMID 24768654
- [Background] Burgos F, Disdier C, de Santamaria EL, Galdiz B, Roger N, Rivera ML, Hervas R, Duran-Tauleria E, Garcia-Aymerich J, Roca J; e-Spir@p Group. Telemedicine enhances quality of forced spirometry in primary care. Eur Respir J. 2012 Jun;39(6):1313-8. doi: 10.1183/09031936.00168010. Epub 2011 Nov 10. PMID 22075488
- [Background] Salas T, Rubies C, Gallego C, Munoz P, Burgos F, Escarrabill J. Technical requirements of spirometers in the strategy for guaranteeing the access to quality spirometry. Arch Bronconeumol. 2011 Sep;47(9):466-9. doi: 10.1016/j.arbres.2011.06.005. Epub 2011 Aug 6. English, Spanish. PMID 21821333
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Vargas C, Burgos F, Cano I, Blanco I, Caminal P, Escarrabill J, Gallego C, Llauger MA, Miralles F, Solans O, Vallverdu M, Velickovski F, Roca J. Protocol for regional implementation of collaborative lung function testing. NPJ Prim Care Respir Med. 2016 Jun 2;26:16024. doi: 10.1038/npjpcrm.2016.24. No abstract available. PMID 27251304